CLINICAL TRIAL: NCT02459158
Title: A Randomized, Open-Label Phase 1b Study of ME1100 Inhalation Solution Plus Best Available Therapy in the Treatment of Mechanically Ventilated Subjects With Bacterial Pneumonia
Brief Title: A Study to Assess the Pharmacokinetic Profile, the Safety, and the Tolerability of ME1100 Inhalation Solution in Patients With Mechanically Ventilated Bacterial Pneumonia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Meiji Seika Pharma Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ME1100-CL-103
Record Dates: First submitted 2015-05-28; First posted 2015-06-01 (Estimated); Last update posted 2017-07-05 (Actual); Status verified 2016-11

CONDITIONS: Pneumonia, Bacterial
MeSH Terms: conditions — Pneumonia, Bacterial

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Low dose of ME1100 (Experimental)
  Interventions: Drug: ME1100 inhalation solution
- High dose of ME1100 (Experimental)
  Interventions: Drug: ME1100 inhalation solution

INTERVENTIONS:
Drug: ME1100 inhalation solution — Low dose of ME1100 inhalation solution twice daily for up to 14 days to be administered via eFlow nebulizer system
  Other Names: Arbekacin inhalation solution
  Arms: Low dose of ME1100
Drug: ME1100 inhalation solution — High dose of ME1100 inhalation solution twice daily for up to 14 days to be administered via eFlow nebulizer system
  Other Names: Arbekacin inhalation solution
  Arms: High dose of ME1100

SUMMARY:
This study is a randomized, open-label phase I study. The primary objective of this study is to assess the pharmacokinetic (PK) profile of ME1100 in subjects with mechanically ventilated bacterial pneumonia (MVBP). The secondary objective of this study is to assess the safety and tolerability of ME1100 for the treatment of subjects with MVBP to assess the safety and tolerability of ME1100.

ELIGIBILITY:
Inclusion Criteria:

Participants must meet all of the following inclusion criteria in order to be eligible for the study:

1. Is a hospitalized male or female, ≥ 18 years of age at the Screening Visit;
2. Is on mechanical ventilation;
3. Has a known or suspected mechanically ventilated bacterial pneumonia with at least 1 of the following:

   * Fever (> 38.5ﾟC or > 101.3ﾟF);
   * Hypothermia (≤ 35.0ﾟC or ≤ 95.0ﾟF);
   * Leukopenia (≤ 4500 cells/mm3);
   * Leukocytosis (≤ 10000 cells/mm3);
   * White blood cell count with left shift defined as > 15% immature polymorphonuclear leukocytes (bands) on peripheral blood smear; or
   * Procalcitonin > 0.25 µg/mL;

   Plus at least 2 of the following:
   * Respiratory failure requiring mechanical ventilation;
   * New onset of expectorated or suctioned purulent sputum production or respiratory secretions, or a change in the character of sputum;
   * Auscultatory findings on pulmonary examination of rales and/or evidence of pulmonary consolidation;
   * Dyspnea, tachypnea, or signs of respiratory distress as evidenced by an increase in respiratory support or oxygen requirement, particularly if any or all of these are progressive in nature; or
   * Hypoxemia by pulse oximetry or arterial blood gas requiring an increase in supplemental oxygen;
4. Has a chest X-ray with a new consolidation consistent with pneumonia or significant worsening of previous findings consistent with pneumonia; and
5. Has an Acute Physiology and Chronic Health Evaluation II (APACHE II) score ≥ 8 and ≤ 30 at the Screening Visit.

Exclusion Criteria:

Participants who meet any of the following exclusion criteria will not be enrolled in the study:

1. Has a requirement of inhaled non-study antibiotic;
2. Has been treated with any inhaled antibiotic (including inhaled aminoglycosides) within 72 hours of study entry;
3. Has renal insufficiency at Screening as evidenced by an estimated creatinine clearance <50 mL/min based on the Cockcroft-Gault formula;
4. Is at risk of rapidly fatal illness and death within the next 72 hours;
5. Is a pregnant or nursing female. Females of childbearing potential must have a serum pregnancy test prior to enrollment. If results of the serum pregnancy test are not available prior to the Day 1 Treatment Visit, the patients may be enrolled on the basis of a negative urine pregnancy test; however, the results of the serum pregnancy test must still be obtained. If either test is positive, the patients must be excluded;
6. Has myasthenia gravis, parkinsonism, or any other progressive neuromuscular disorder;
7. Has a history of epilepsy or known seizure disorder;
8. Has a history of sensorineural hearing loss resulting from any therapy known as ototoxic (eg, aminoglycosides, cisplatin, loop diuretics, or quinine);
9. Has received any investigational medication in the last 30 days (or 5 half-lives of the investigational medication, whichever is longer) prior to the Screening Visit; or
10. Has known hypersensitivity to ME1100, aminoglycosides, or any of the specified Best Available Therapy agents or their excipients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2015-09; Primary Completion 2017-03-22 (Actual); Study Completion 2017-03-22 (Actual)

PRIMARY OUTCOMES:
Arbekacin concentrations in respiratory fluids collected via bronchoalveolar lavage (BAL) for epithelial lining fluid (ELF) | Day 3
Plasma arbekacin concentrations | Day 1 to Day 5
Urinary elimination of arbekacin | Day 2
Arbekacin concentrations in tracheal aspirate | Day 2

SECONDARY OUTCOMES:
Number of participants with adverse events | Screening through 14 days after the end of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Meiji Study Director, Study Director — Meiji Seika Pharma Co., Ltd.
Locations (14):
- United States (14):
  - Martinez, California
  - Sacramento, California
  - San Diego, California
  - Aurora, Colorado
  - Jacksonville, Florida
  - Hazard, Kentucky
  - Worcester, Massachusetts
  - Kalamazoo, Michigan
  - Buffalo, New York
  - Greensboro, North Carolina
  - Cincinnati, Ohio
  - Lima, Ohio
  - Toledo, Ohio
  - Houston, Texas